CLINICAL TRIAL: NCT05636358
Title: Hypnotherapy Through Self-exercises in Children With Functional Abdominal Pain in Primary Care
Acronym: ZelfHy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL73562.042.20; NL8500 (Registry Identifier: Dutch Trial Register); 852002035 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-11-14; First posted 2022-12-05 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Functional Gastrointestinal Disorders; Irritable Bowel Syndrome; Functional Abdominal Pain Syndrome
Keywords: Primary care; Children and adolescents
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This study is a pragmatic randomised controlled trial (RCT) with a total follow-up of 12 months executed in primary care in the Netherlands. Participating children will be randomised 1:1 on the patient level to either the intervention or the care as usual group. The intervention group will receive 3 months home-based hypnotherapy by self-exercises in addition to care as usual by their GPs according to the Dutch Society of GPs' (NHG) guideline. The control group will receive usual care (UC) by their GPs alone according to the Dutch Society of GPs' (NHG) guideline.
Who Masked: Outcomes Assessor
Masking Description: Although the children and GP's cannot be blinded to the allocation, researchers performing the analyses will be blinded for allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based hypnotherapy (Experimental): The intervention includes existing home-based hypnotherapy self-exercises in MP3 format for a period of three months.
  The intervention group of children with FAP or IBS in primary care receives the home-based hypnotherapy self exercises in addition to care as usual by their GP according to the guideline commissioned by the Dutch Society of GPs.
  Interventions: Other: Home-based hypnotherapy
- Control (No Intervention): The control group of children with FAP or IBS in primary care will receive only care as usual by their GP. After the end of the study, the control group will also receive access to the home-based hypnotherapy exercises, if desired.

INTERVENTIONS:
Other: Home-based hypnotherapy — The home-based hypnotherapy package contains five standard hypnosis exercises. They consist of one breathing exercise, and four visualisation exercises. Two separate sets adjusted to the child's age will be used: one for children younger than 12 years and one for children of 12 years and older. The children will be asked to listen to the exercises at least 5 times per week, for approximately 15-20 minutes per day, during a period of 3 months. A workbook will provide children and/or parents with the instructions and planning of the exercises.
  Arms: Home-based hypnotherapy

SUMMARY:
The goal of this randomised controlled trial is to study the (cost-)effectiveness of home-based hypnotherapy by self-exercises in children with functional abdominal pain (FAP) or irritable bowel syndrome (IBS) in primary care. The main questions it aims to answer are:

* What is the effect of home-based hypnotherapy by self-exercises on adequate relief of abdominal pain and discomfort in addition to care as usual of general practitioners (GPs), compared to care as usual of GPs alone in children with FAP or IBS?
* What is the effect of home-based hypnotherapy by self-exercises in addition to care as usual by GPs compared to care as usual of GPs alone in children with FAP or IBS on:

  * Frequency and intensity of abdominal pain and discomfort
  * Pain severity
  * Daily functioning and impact
  * Anxiety and depression
  * Pain beliefs
  * Sleep disturbances
  * School absence
  * Use of health care services, including GP visits and referrals to secondary care
  * Costs (healthcare and societal perspective)

Participants in the intervention group will receive home-based hypnotherapy 5 times a week for approximately 15-20 minutes a day during 3 months in addition to care as usual by their GP according to the Dutch society of GPs' guideline for children with abdominal pain.

Participants in the control group will receive care as usual by their GP according to the Dutch society of GPs' guideline for children with abdominal pain.

DETAILED DESCRIPTION:
Recruitment

This study will be performed within the network of GPs connected to the Department of General Practice of the UMCG (Academisch Huisarts Ontwikkel Netwerk, AHON).

Children and/or parents visiting the GP with chronic gastrointestinal symptoms (at least 4 days per month during the past 2 months), who had none of the exclusion criteria, will be approached by their general practitioner (GP), either during consultation or following monthly retrospective search of medical records. The GP fills out the study response form including the in- and exclusion criteria and the contact details of the child and/or parents. If the child seems eligible, the child and/or parents will receive the patient information letter. If the child and/or parents are interested in study participation and provide permission, the GP will send the response form to the research team.

To further improve patient recruitment, since August 2022 children and parents are informed through schools, (social) media and the study website. Information includes background on functional abdominal pain (FAP) and irritable bowel syndrome (IBS), hypnotherapy, the current study, and contact information of the research group. The researchers will contact children and/or parents who apply for participation by telephone. The researcher will answer questions and check eligibility criteria. If the child wishes to participate, the researcher sends the PIF and informed consent (IC) forms via a REDCap link to their e-mail address. In the same e-mail, the researcher informs how their GP can find information and the digital response form on the study website. The GP will check the in- and exclusion criteria prior to participation and directly submits the form to the researchers on the study website.

The researcher/research assistant will approach the eligible children and/or parents by telephone within one week after receiving their response form. During the call the researcher/research assistant fills out the Rome IV criteria questionnaire and checks whether the child and/or parents are motivated and willing to participate. Questions by the child and/or parents will be answered. If the child is willing to participate, the researcher/research assistant will inform the child and/or parents, and send the IC forms via a REDCap link to their e-mail address to those who were included directly during consultation. If preferred, the second contact moment may also be face-to-face in the GP's practice instead. A follow-up visit at the GP 4 weeks after inclusion should also be scheduled. If the child does not want to be randomised, the child and/or parents are asked whether they are willing to participate in a cohort. Here, children with chronic abdominal pain and their parents will not participate in the RCT, but they will fill out primary and secondary parameters like in the RCT at baseline and during follow-up via the online system REDCap. If they are willing to participate in the cohort, they will also receive IC forms to be signed via REDCap. The research team will continuously monitor the return of the IC forms, and will call the child and/or parents if they do not return the forms. If child and/or parent(s) prefer written information and IC, the patient information package including a return envelope can be sent by regular post.

After signing the digital IC forms in REDCap, all children and/or parents will be asked to fill-out the baseline parameters online via a digital link from REDCap. They cannot begin with the questionnaires before giving informed consent. Next, randomisation will be performed. The result from the randomisation procedure will be discussed during the second telephone call by the research team and the child and/or parents. During this call the researcher/research assistant will also inform the IG about intervention procedures. The workbook in the online portal is leading and self-explanatory. Questions will be answered. Afterwards, the intervention group (IG) will receive access to the home-based hypnotherapy self-exercises for 3 months via a login to the closed part of the website/portal. All children in both the RCT and the cohort will fill out the required primary and secondary parameters at baseline, 3, 6 and 12 months through the digital REDCap application.

Overall, the GP remains responsible for the medical health of the children and will respond to any medical issues or related questions. The researchers are responsible for guiding the practical questions in relation to the study. To help the child and/or parents with practical issues, the public part of the website/portal contains a section on frequently asked questions (FAQ).

Statistical analysis In general, the researchers will use appropriate descriptive statistics and frequencies to summarize the collected primary and secondary outcomes at baseline and during follow-up.

Primary study outcomes

The primary outcome is the proportion of children with self-identified adequate relief of abdominal pain/discomfort (yes/no) after 12 months follow-up in the intervention group versus the care as usual group. The researchers will perform an intention to treat in a primary analysis and per protocol in a secondary analysis. The intention to treat population includes all children with signed IC, who have been randomised (despite what treatment they have in fact received). The per protocol population includes the children, who in fact have had the home-based hypnotherapy self-exercises and the control group, who in fact had no home-based hypnotherapy self-exercises.

A missing value analysis will be performed and if missing values are more than 5% and considered missing at random (MAR), data will be imputed by multiple imputation. The primary outcome is analyzed with an intention-to-treat analysis using a multivariable logistic regression model. Covariates taken into consideration include the stratification factor based upon age (<12 years versus ≥12 years), baseline pain severity score (NRS-11) and treatment expectations of the child and parents at baseline. Both a complete cases analysis and an analysis with the imputed data (if the missing data are considered MAR) will be performed. A secondary per protocol analysis of the responders in the IG will be performed based on adequate use of the intervention. Adequate use is defined as listening to one of the exercises for at least 80% of the time.

Secondary study outcomes

The researchers will use logistic and linear multilevel analyses to investigate the longitudinal relationship between the intervention group and the control group with respect to the various secondary outcome variables. This includes the frequency and intensity of the abdominal pain/discomfort, school absence, anxiety and depression, pain beliefs, functional impairment and impact, sleep scores and healthcare use. The applied levels will be the repeated measures (the time - baseline, 3 months, 6 months and 12 months) and the patient groups respectively.

The cost effectiveness will be measured with a time horizon of 12 months, and costs will be calculated from a societal perspective. The cost-effectiveness analysis will include the primary outcome, expressing the additional costs or savings per additional patient with adequate relief of symptoms. Data regarding health care consumption and productivity losses will be collected on a patient level. Cost categories to be included are for example costs of the online intervention application, GP and specialist visits, medication, and productivity losses of parents. The cost questionnaire and the medical records of the participating child will be used to collect data regarding health care consumption and productivity losses. These items will be valued using standard prices from the Zorginstituut and medicijnkosten.nl when possible. For the use of the online intervention application, a cost price will be calculated based on true resources used. Costs between the two treatment arms will be compared. In the cost utility analysis, patient outcome will be measured using the EuroQoL Youth (EQ-5D-Y) and compared per study group.

Other study parameters

Patient descriptive data, Rome IV criteria, treatment expectations, frequency and intensity of the use of the hypnotherapy self-exercises and co-morbid somatization problems will be presented with the appropriate descriptive statistics and frequencies to summarize the information. School level and treatment expectations will be incorporated as covariates in the analyses of the primary outcome. Usage of the hypnotherapy self-exercises will be integrated in the responder analysis of the intervention group.

Sample size calculation

Based on earlier research, the researchers expect adequate relief in 55% of the children in the usual care group and 75% in the intervention group. In order to detect this difference of 20%, with 80% power and 5% significance level a randomised study would require 180 children (90 per group). When taking into account a total loss during follow-up of 10%, the researchers need to include 200 children (100 per group) for this study.

Handling and storage of data and documents

All consecutive patients, who meet the inclusion criteria, will receive a unique study number, assigned by the coordinating investigator. The study number is not based on the patient's initials and birth-data. The study number will be composed of the number of inclusion and the stratification group (<12 years or ≥12 years). All data will be collected and stored linked to this number. All patients, who gave written IC for the study, will complete digital questionnaires via a hyperlink to REDCap send by e-mail, which will automatically be linked to the corresponding study ID. The coordinator investigator has access to the full subject identification code lists in order to able to link patients to the corresponding study number. A password is needed for entering this link file. Data will be stored during the study period and until 15 years thereafter when the parents give permission.

Monitoring and quality assurance

As this study is with negligible risks a monitor from the UMCG Monitor pool will monitor the study once 50 participants are recruited. A qualified monitor (research assistant at the Department of General Practice and Elderly Care Medicine, UMCG) has prepared a concept monitoring plan, including specification of the methods, frequency and extent of the monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7 to 17 years
* GP visit concerning chronic gastrointestinal symptoms
* FAP or IBS according to their GP

Exclusion Criteria:

* A concomitant organic gastrointestinal disease
* Treatment by a paediatrician for abdominal symptoms
* Intellectual disability
* A history of a psychotic disorder
* Hypnotherapy treatment in the past year
* Insufficient knowledge of the Dutch language by the child or parents

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Adequate relief at 12 months | 12 months
  Proportion of children with adequate relief of abdominal pain at 12 months follow-up Child and/or parents are asked whether the child has adequate relief of FAP or IBS related abdominal pain during the past week using a dichotomous scale (yes/no). This question is a well validated outcome measurement in trials on treatment for IBS.

SECONDARY OUTCOMES:
Adequate relief at 3 and 6 months | 3 and 6 months
  Proportion of children with adequate relief of abdominal pain at 3 and 6 months follow-up Child and/or parents are asked whether the child has adequate relief of FAP or IBS related abdominal pain during the past week using a dichotomous scale (yes/no). This question is a well validated outcome measurement in trials on treatment for IBS.
Pain frequency and intensity | 0, 3, 6, and 12 months
  Child and/or parents will assess the abdominal pain or discomfort during seven consecutive days with a diary at baseline and during follow-up. A score of seven days is totalled in a pain frequency score (range 0 tot 21) and a pain intensity score (range 0 to 21). A reduction in abdominal pain/discomfort is defined as at least 50% reduction in both scores.
Severity of pain | 0, 3, 6, and 12 months
  Child and/or parents will assess the severity of the abdominal pain or discomfort during the past week with a 0-10 numerical rating scale (NRS-11) at baseline and during follow-up. The NRS-11 is also integrated as outcome measure for pain/discomfort, because there is much heterogeneity between various pain scales. This scale measures pain severity, while the pain diary reports also frequency, intensity and duration of the pain and/or discomfort in order to complement each other.
Daily functioning and impact | 0, 3, 6, and 12 months
  Child and/or parents will assess the impact of the abdominal pain and discomfort on their daily functioning and quality of life with the KIDSCREEN-52. The KIDSCREEN-52 is a health-related quality of life questionnaire for children and adolescents. It includes 52 items covering ten dimensions of physical, psychologic and social aspects. The instrument has sound measurement properties and is available in Dutch.
Anxiety and depression | 0, 3, 6, and 12 months
  Child and/or parents will assess their mental well-being using the short version of the Revised Child Anxiety and Depression Scale (RCADS-25). Children will be asked to indicate how often each item (15 anxiety items and 10 depression items) applies to them according to a 4-point scale (never to always) at baseline and during follow-up. The validity and reliability for both subscales of this short version of the RCADS were acceptable and not significantly different from the extensive version of the RCADS.
Pain beliefs | 0, 3, 6, and 12 months
  Child and/or parents will score the pain beliefs with the paediatric Pain Beliefs Questionnaire (PBQ) at baseline and during follow-up. This questionnaire consists of 32 items scored on a 5-point Likert scale.
Sleep disturbances | 0, 3, 6, and 12 months
  Child and/or parents will evaluate sleep disturbances with three selected questions from the validated Sleep Self Report: 1) Do you fall asleep in about 20 minutes? 2) Do you wake up at night when your parents think you are asleep? 3) Do you feel sleepy during the day? Children will be asked to indicate the frequency of occurrence of these items in the past week in three categories: rarely (0-1 time per week), sometimes (2-4 times per week), and usually (5-7 times per week).
School absence | 0, 3, 6, and 12 months
  Parents will administer the missed days at school during the past 3 months prior to baseline and during follow-up. The question is integrated in the cost-questionnaire administered to parents.
Healthcare consumption | 0, 3, 6, and 12 months
  Medical records of the participating children will be screened at 12-months follow-up by the researcher/research assistant for the number of GP visits due to functional somatic symptoms and/or FAP or IBS; referrals due to FAP or IBS; and medication use over the past year.
Cost-effectiveness | 0, 3, 6, and 12 months
  The cost-effectiveness analysis will be based upon the iMTA instruments (productivity cost questionnaire and medical consumption questionnaire) to collect data regarding health care consumption and productivity losses.
Cost-utility | 0, 3, 6, and 12 months
  For the cost-utility analysis, child and/or parents will score the EuroQoL Youth (EQ-5D-Y), which is a generic measure for quality of life suitable for utility calculations. This instrument includes five items (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and three levels of severity problems (no problems, some problems, a lot of problems). The questionnaire is feasible, reliable and valid, and developed for children aged 8 years and older.

OTHER OUTCOMES:
Patient baseline characteristics | Baseline
  Patient baseline characteristics will be collected from the GP's inclusion form / response card include gender, age/birthdate, and school level. Data on co-morbidities/medical history and medication use will be extracted from the child's medical records at the GP's practice after 12 months follow-up.
Paediatric gastrointestinal symptoms | Baseline
  Paediatric gastrointestinal symptoms at baseline are measured using the Dutch version of the Rome IV questionnaire. The Rome IV consists of a parent report, and a self-report for children aged 10 years and older.
Usage of hypnotherapy self-exercises | 3 months
  Data on the frequency and duration of the intervention use as well as the exercises selected will be obtained from the online website/portal for the IG only after the 3 months intervention period.
Treatment expectations | Baseline
  To evaluate placebo effects, one question will be incorporated at baseline about whether the child and parents (asked separately) expect that the symptoms will improve with the treatment on an 11-point scale (0 = not at all; 10 = complete recovery). They will also be asked whether they have a preference for the IG or the CG.
Quality of exercises | 3 months
  Each exercise will be rated with an overall score (range 0 - 10) as well as qualitatively by asking to fill out positives and negatives. This will be done after 3 months for the IG only.
Somatisation | 0, 3, 6, and 12 months
  Child and/or parents will evaluate the experienced somatic symptoms by scoring the Children's Somatization Inventory (CSI). The inventory consists of 35 items on physical symptoms with a scoring scale per item ranging from 0 (no problems at all) to 4 (a whole lot). A total score can be computed by summing the scores across all items, with higher scores indicating a higher intensity of functional complaints. The inventory has been translated into Dutch and has good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Y. Berger, prof, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
(Several versions of) processed data, syntaxes, data documentation and raw data will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After all publications concerning the study are published.
Access Criteria: Data will be made available upon reasonable request.

REFERENCES:
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632
- [Background] Rutten JMTM, Vlieger AM, Frankenhuis C, George EK, Groeneweg M, Norbruis OF, Tjon A Ten W, van Wering HM, Dijkgraaf MGW, Merkus MP, Benninga MA. Home-Based Hypnotherapy Self-exercises vs Individual Hypnotherapy With a Therapist for Treatment of Pediatric Irritable Bowel Syndrome, Functional Abdominal Pain, or Functional Abdominal Pain Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2017 May 1;171(5):470-477. doi: 10.1001/jamapediatrics.2017.0091. PMID 28346581
- [Background] Lisman-van Leeuwen Y, Spee LA, Benninga MA, Bierma-Zeinstra SM, Berger MY. Prognosis of abdominal pain in children in primary care--a prospective cohort study. Ann Fam Med. 2013 May-Jun;11(3):238-44. doi: 10.1370/afm.1490. PMID 23690323
- [Background] Gieteling M, Van Dijk P, De Jonge A, Albeda F, Berger M, Burgers J. NHG-Standaard Buikpijn bij kinderen. Huisarts Wet 2012; 55: 404-409.
- [Background] Mangel AW, Hahn BA, Heath AT, Northcutt AR, Kong S, Dukes GE, McSorley D. Adequate relief as an endpoint in clinical trials in irritable bowel syndrome. J Int Med Res. 1998 Mar-Apr;26(2):76-81. doi: 10.1177/030006059802600203. PMID 9602985
- [Background] Saps M, van Tilburg MA, Lavigne JV, Miranda A, Benninga MA, Taminiau JA, Di Lorenzo C. Recommendations for pharmacological clinical trials in children with irritable bowel syndrome: the Rome foundation pediatric subcommittee on clinical trials. Neurogastroenterol Motil. 2016 Nov;28(11):1619-1631. doi: 10.1111/nmo.12896. Epub 2016 Jul 31. PMID 27477090
- [Background] Castarlenas E, Jensen MP, von Baeyer CL, Miro J. Psychometric Properties of the Numerical Rating Scale to Assess Self-Reported Pain Intensity in Children and Adolescents: A Systematic Review. Clin J Pain. 2017 Apr;33(4):376-383. doi: 10.1097/AJP.0000000000000406. PMID 27518484
- [Background] Ravens-Sieberer U, Gosch A, Rajmil L, Erhart M, Bruil J, Duer W, Auquier P, Power M, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J, Kidscreen Group E. KIDSCREEN-52 quality-of-life measure for children and adolescents. Expert Rev Pharmacoecon Outcomes Res. 2005 Jun;5(3):353-64. doi: 10.1586/14737167.5.3.353. PMID 19807604
- [Background] Ebesutani C, Reise SP, Chorpita BF, Ale C, Regan J, Young J, Higa-McMillan C, Weisz JR. The Revised Child Anxiety and Depression Scale-Short Version: scale reduction via exploratory bifactor modeling of the broad anxiety factor. Psychol Assess. 2012 Dec;24(4):833-45. doi: 10.1037/a0027283. Epub 2012 Feb 13. PMID 22329531
- [Background] Stone AL, Walker LS, Laird KT, Shirkey KC, Smith CA. Pediatric Pain Beliefs Questionnaire: Psychometric Properties of the Short Form. J Pain. 2016 Sep;17(9):1036-44. doi: 10.1016/j.jpain.2016.06.006. Epub 2016 Jun 27. PMID 27363626
- [Background] Steur LMH, Grootenhuis MA, Terwee CB, Pillen S, Wolters NGJ, Kaspers GJL, van Litsenburg RRL. Psychometric properties and norm scores of the sleep self report in Dutch children. Health Qual Life Outcomes. 2019 Jan 16;17(1):15. doi: 10.1186/s12955-018-1073-x. PMID 30651118
- [Background] iMTA Productivity Cost Questionnaire and iMTA Medical Consumption Questionnaire. Retrieved at the 9th of April 2020 from https://www.imta.nl/questionnaires/.
- [Background] Wille N, Badia X, Bonsel G, Burstrom K, Cavrini G, Devlin N, Egmar AC, Greiner W, Gusi N, Herdman M, Jelsma J, Kind P, Scalone L, Ravens-Sieberer U. Development of the EQ-5D-Y: a child-friendly version of the EQ-5D. Qual Life Res. 2010 Aug;19(6):875-86. doi: 10.1007/s11136-010-9648-y. Epub 2010 Apr 20. PMID 20405245
- [Background] Ravens-Sieberer U, Wille N, Badia X, Bonsel G, Burstrom K, Cavrini G, Devlin N, Egmar AC, Gusi N, Herdman M, Jelsma J, Kind P, Olivares PR, Scalone L, Greiner W. Feasibility, reliability, and validity of the EQ-5D-Y: results from a multinational study. Qual Life Res. 2010 Aug;19(6):887-97. doi: 10.1007/s11136-010-9649-x. Epub 2010 Apr 17. PMID 20401552
- [Background] Rutten JM, Vlieger AM, Frankenhuis C, George EK, Groeneweg M, Norbruis OF, Tjon a Ten W, Van Wering H, Dijkgraaf MG, Merkus MP, Benninga MA. Gut-directed hypnotherapy in children with irritable bowel syndrome or functional abdominal pain (syndrome): a randomized controlled trial on self exercises at home using CD versus individual therapy by qualified therapists. BMC Pediatr. 2014 Jun 4;14:140. doi: 10.1186/1471-2431-14-140. PMID 24894077
- [Background] Meesters C, Muris P, Ghys A, Reumerman T, Rooijmans M. The Children's Somatization Inventory: further evidence for its reliability and validity in a pediatric and a community sample of Dutch children and adolescents. J Pediatr Psychol. 2003 Sep;28(6):413-22. doi: 10.1093/jpepsy/jsg031. PMID 12904453
- [Derived] Ganzevoort IN, Berger MY, Vlieger AM, Benninga MA, De Boer MR, Holtman GA. Children with disorders of gut-brain interaction in primary care versus hospital care: A comparison of characteristics. J Pediatr Gastroenterol Nutr. 2025 Sep;81(3):530-539. doi: 10.1002/jpn3.70129. Epub 2025 Jun 29. PMID 40581866
- [Derived] Ganzevoort IN, Fokkema T, Mol-Alma HJ, Heida A, Van der Veen AL, Vermeulen K, Benninga MA, Vlieger AM, Berger MY, Holtman GA. Home-based guided hypnotherapy for children with functional abdominal pain and irritable bowel syndrome in primary care: study protocol for a randomised controlled trial. BMJ Open. 2023 May 8;13(5):e069653. doi: 10.1136/bmjopen-2022-069653. PMID 37156587